CLINICAL TRIAL: NCT04692714
Title: Evaluation of Two Surgical Strategies for Robotic Implantation of Total Knee Prostheses (Stryker), Cemented Versus Uncemented. Prospective, Randomized, Single-center, Multisite Non-inferiority Study.
Brief Title: Evaluation of Two Surgical Strategies for Robotic Implantation of Total Knee Prostheses (Stryker), Cemented Versus Uncemented
Acronym: MAKO CIMENT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: Stryker Nordic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 69HCL20_0872
Record Dates: First submitted 2020-12-30; First posted 2021-01-05 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Total Knee Arthroplasty
Keywords: total knee arthroplasty; prosthesis; cement; MAKO; IKS score

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental knee prosthesis implantation (Experimental): Patients included in this arm will have a total knee arthroplasty using a Triathlon prosthesis by STRYKER implemented without additional cement using the MAKO robot
  Interventions: Device: Knee prosthesis implementation without additional cement
- Conventional knee prosthesis implantation (Active Comparator): Patients included in this arm will have a total knee arthroplasty using a Triathlon prosthesis by STRYKER implemented with additional cement using the MAKO robot
  Interventions: Device: Knee prosthesis implementation with additional cement

INTERVENTIONS:
Device: Knee prosthesis implementation with additional cement — During surgery, a TRIATHLON prosthesis will be implemented with the MAKO robot with additional cement.
  Arms: Conventional knee prosthesis implantation
Device: Knee prosthesis implementation without additional cement — During surgery, a TRIATHLON prosthesis will be implemented with the MAKO robot without additional cement.
  Arms: Experimental knee prosthesis implantation

SUMMARY:
Total knee replacement surgery (TKA) is a treatment for advanced tibial-femoral osteoarthritis. This intervention is justified in case of significant discomfort and failure of medical treatment. It aims to replace the native internal and external femoro-tibial joints with a joint between a femoral implant and a tibial implant.

Implants can be cemented or cementless. The longevity of these implants depends among other things on the quality of the bone fixation of the implants. It is therefore essential that this fixation be evaluated. The advantages of an uncemented TKA are the preservation of bone stock, the absence of wear by cement debris and prolonged fixation thanks to osseointegration. These characteristics are all the more interesting in a young population.

Numerous studies have been carried out on the survival of TKA with and without cement. The results found are not unanimous and mainly concern the survival of the implants and the presence of radiological signs of loosening. In addition, no study has evaluated the results of TKA with or without cement implanted using robotic assistance. The precision provided by the robotic system could improve the results of these uncemented implants.

Very few studies are interested in the functional results according to the cementation or not of TKA. And most of these studies do not have a high level of methodological evidence.

We would like to prospectively evaluate the functional results, survival, as well as the rate of radiological border after TKA with or without cement posed with robotic assistance, in the short and medium term.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of internal, external or global femorotibial knee osteoarthritis
* Indication for first-line total knee arthroplasty
* having given informed consent
* Affiliated with a social security scheme
* Patient being able to understand the objectives of the study and willing to comply with postoperative instructions.

Exclusion Criteria:

* Patient with rheumatoid arthritis
* Preoperative flexion less than 90 °
* Prosthesis associated with an osteotomy
* History of surgery on the operated knee, except arthroscopy
* Poor bone quality assessed by the surgeon
* Knee deformation greater than 10 ° preoperatively (HKA)
* Pregnant or breastfeeding Women
* Persons deprived of their liberty by a judicial or administrative decision, persons under psychiatric care, persons admitted to a health or social institution for purposes other than research
* Adults subject to a legal protection measure
* Patient already participating to another clinical trial that might jeopardize the current trial

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-05-16 (Actual); Primary Completion 2025-05-16 (Estimated); Study Completion 2028-10-16 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in International Knee Society (IKS) function score at 12 Months | Baseline and 12 months
  The knee function will be evaluated using the delta of the IKS function score between baseline (before surgery) and 1 year after total knee arthroplasty, and compared between the 2 arms.

SECONDARY OUTCOMES:
Change from baseline in IKS objective score at 12 Months | Baseline and 12 months
  The knee function will be evaluated using the delta of the IKS objective score between baseline (before surgery) and 1 year after total knee arthroplasty, and compared between the 2 arms.
Change from baseline in IKS function score at 60 Months | Baseline and 60 months
  The knee function will be evaluated using the delta of the IKS function score between baseline (before surgery) and 5 years after total knee arthroplasty.
Change from baseline in IKS objective score at 60 Months | Baseline and 60 months
  The knee function will be evaluated using the delta of the IKS objective score between baseline (before surgery) and 5 years after total knee arthroplasty.
Forgotten joint score at 12 Months | 12 months
  Patient prosthesis acceptability will be evaluated thanks to the forgotten joint score 12 months after total knee arthroplasty
Forgotten joint score at 60 Months | 60 months
  Patient prosthesis acceptability will be evaluated thanks to the forgotten joint score 60 months after total knee arthroplasty
Presence of progressive radiological border at 12 Months | 12 months
  Progressive radiological border will be judged significant if it is at least 2 mm long at the interface between the implant (or cement) and the bone, or if it progresses in comparison to immediate post-surgical time.
Unsealing free survival at 60 months | 60 months
  Unsealing free survival of knee prosthesis 60 months after total knee arthroplasty

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien LUSTIG, Professor, Principal Investigator — Hospices Civils de Lyon
Locations (2):
- France (2):
  - Department of orthopedic surgery, Hopital Nord Croix-Rousse- Hospices Civils de Lyon, Lyon
  - Chirurgie Orthopédique et Traumatologique Centre Hospitalier Lyon Sud, Hospices Civils de Lyon, Lyon

REFERENCES:
- See also: Related Info — http://www.orthopedie-lyon-croix-rousse.fr/equipe-chirurgien-orthopediste-lyon-69.html